CLINICAL TRIAL: NCT03555812
Title: Pelvic Inclination Measurement by Navigated Ultrasound
Acronym: MIPEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29BRC18.0061 MIPEN
Record Dates: First submitted 2018-05-14; First posted 2018-06-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2019-08

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Hip, Arthroplasty, pelvic inclination, ultrasound

STUDY DESIGN:
Intervention Model Description: measurements of pelvic inclination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Experimental): * a medical examination
  * 10 measurements of pelvic tilt in sitting position, 10 measurements of pelvic tilt in supine position and 10 measurements of pelvic tilt in standing position, each performed by three different operators. These measurements will be done by ultrasound.
  Interventions: Other: Pelvic inclination measurement
- Patients (Experimental): a consultation the day before surgery, and a consultation 2 months after surgery, each including:
  * a medical examination
  * 3 pelvic tilt measurements (1 standing, 1 sitting and 1 lying down). These measurements will be done by ultrasound.
  Interventions: Other: Pelvic inclination measurement

INTERVENTIONS:
Other: Pelvic inclination measurement — Measurement of pelvic inclination per ultrasound

SUMMARY:
Prospective, multicenter, non-randomized study.

Primary endpoint : to confirm the proper functioning of the device in vivo by analyzing intra and interobserver reproducibility of repeated measurements on healthy controls.

Secondary endpoint : to describe the values of pelvic inclination while standing, sitting and lying in patients with severe hip osteoarthritis before and after total hip arthroplasty

After signing the inform consent form:

For the first endpoint (, 3 healthy volunteers of different morphotypes will have one consultation comprising :

* a medical examination
* 10 measurements of pelvic inclination in sitting position, 10 measurements of pelvic inclination in supine position and 10 measurements of pelvic inclination in standing position, each realized per three different operators. These measurements will be carried out with navigated ultrasound.

For the secondary endpoint, 30 patients awaiting for a hip replacement surgical intervention will realized one consultation the day before the intervention, and one consultation at 2 months after surgery, each comprising :

* a medical examination
* 3 measurements of pelvic inclination (1 standing, 1 sitting and 1 supine). These measurements will be carried out with navigated ultrasound.

ELIGIBILITY:
Inclusion Criteria:

For primary endpoint

* No medical or surgical history
* Major healthy voluntary topic with

  * Body Mass Index (BMI) <20 for a subject
  * 24 <BMI <26 for a subject
  * BMI> 30 for a subject
* Subject having signed an informed consent

For the secondary endpoint

* Adult patient requiring total hip arthroplasty for severe hip osteoarthritis
* Patient having signed an informed consent

Exclusion Criteria:

* Minor subject
* Resumption of total hip prosthesis
* Subject who can not express their consent to research
* Presence of medical or surgical history for healthy volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Pelvic inclination measurement | Day 0
  The pelvic inclination measurement corresponds to the anterior pelvic plane also known as the Lewinnek's plane; defined by the plane between both anterior superior iliac spine and the pubic symphysis.
  A Portable Ultrasound based Device is used for the Measurement of the Pelvic Tilt

SECONDARY OUTCOMES:
Variation of pelvic inclination before and after hip replacement | Month 2
  The pelvic inclination measurement corresponds to the anterior pelvic plane also known as the Lewinnek's plane; defined by the plane between both anterior superior iliac spine and the pubic symphysis.
  A Portable Ultrasound based Device is used for the Measurement of the Pelvic Tilt

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique de Keraudren, Brest
  - Brest University Hospital, Brest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dardenne G, Pluchon JP, Letissier H, Guezou-Philippe A, Gerard R, Lefevre C, Stindel E. Accuracy and Precision of an Ultrasound-Based Device to Measure the Pelvic Tilt in Several Positions. J Ultrasound Med. 2020 Apr;39(4):667-674. doi: 10.1002/jum.15141. Epub 2019 Oct 30. PMID 31665548